CLINICAL TRIAL: NCT06668168
Title: The Causal Role of Ketone Bodies in Obesity-Associated Disease Prevention - Combining Genetic Epidemiology With a Randomised Trial to Infer Causality
Acronym: KETO-GENETIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: University of Bristol (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Professor of Nutrition and Metabolism, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23-09665
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Nutrition; Obesity and Overweight
Keywords: Ketogenic diet
MeSH Terms: conditions — Obesity; Overweight | interventions — Diet, Ketogenic

STUDY DESIGN:
Masking Description: Outcome assessors will be masked to the group allocation when analysis is outsourced from the University.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (No Intervention)
- KETONE ESTER (Active Comparator)
  Interventions: Dietary Supplement: Ketone Monoester (KE)
- KETOGENIC DIET (Experimental)
  Interventions: Behavioral: Ketogenic diet

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KE) — 25g ketone ester 3x/day. The ketone ester will be a beta-hydroxybutyrate monoester [(R)-3-hydroxybutyl (R)-3-hydroxybutyrate].
  Arms: KETONE ESTER
Behavioral: Ketogenic diet — Ketogenic diet (<50 g carbohydrate per day)
  Arms: KETOGENIC DIET

SUMMARY:
Excess weight increases the risk of several diseases including cardiovascular disease, type 2 diabetes, kidney disease and various cancers. There is a need for preventative strategies for obesity-associated disease, especially for people in the overweight and moderately obese ranges where pharmacological intervention may not be suitable.

Low-carbohydrate (ketogenic) diets are popular for weight control. Ketogenic diets increase circulating ketones, which can have favourable effects on cardiometabolic health markers. However, the ketogenic diet has a nutrient composition associated with harms (high-saturated fat/red meat, and low-fibre). The net effects of ketogenic diets on long-term health are unclear. Ketone supplements can increase circulating ketones and could provide benefits of ketosis without needing to adhere to a potentially harmful diet.

Establishing causality between complex exposures (e.g., diet) and long-term outcomes (e.g., disease), is challenging. The MRC & NIHR Review of Nutrition and Human Health Research (2017) highlighted an "overreliance (as opposed to reasonable reliance) on observational studies" as a key barrier to progression in the field of nutrition and health. Randomised controlled trials (RCTs) facilitate causal inference, but for long-term outcomes are expensive, time-consuming, and often suffer from waning adherence. Mendelian randomization (MR) can estimate causal effects subject to key assumptions. A challenge to these assumptions includes complex behavioural exposures (e.g., diet), which could be intercorrelated with causal factors.

Our proposal will address these limitations with a novel combination of study designs to establish causal effects of ketosis (via diet and supplementation) on obesity-associated disease risk in humans.

The investigators will combine a tightly controlled, short-term RCT, with MR to link short-term responses to long-term endpoints. The investigators will examine the circulating (blood) and tissue-specific (adipose) transcriptomic and proteomic responses in the fasted and postprandial state in response to our dietary interventions and translate these to MR by identifying single-nucleotide polymorphisms from genome wide association studies. This approach overcomes limitations of RCTs and MR, as adherence to diets will be confirmed with controlled feeding, and intermediate molecular traits as exposure for MR are less likely to be intercorrelated with causal traits.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index: 25-45 kg/m2
* Waist circumference >93.9 (males) or >79.9 (females)

Exclusion Criteria:

* Glucose or lipid lowering medication
* Diagnosis of cardiovascular disease, renal failure, liver disease or type 2 diabetes
* Contraindications to a ketogenic diet (e.g., pancreatitis, liver failure, disorders of fat metabolism, primary carnitine deficiency, carnitine palmitoyltransferase deficiency, carnitine translocase deficiency, porphyrias, or pyruvate kinase deficiency)
* Unable to understand English language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-05-06 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Plasma proteome | From baseline to week 4
  Plasma proteome at week 4 adjusted for baseline values
Transcriptome of peripheral blood mononuclear cells | From baseline to week 4
  Transcriptome of peripheral blood mononuclear cells at week 4 adjusting for baseline values
Transcriptome of adipose tissue | From baseline to week 4
  Transcriptome of subcutaneous abdominal adipose tissue at week 4 adjusting for baseline values

SECONDARY OUTCOMES:
Apolipoprotein B concentrations | From baseline to week 4
  Plasma apolipoprotein B concentrations at week 4 adjusted for baseline values.
Urinary albumin concentrations | From baseline to week 4
  Urinary albumin concentrations at week 4 adjusting for baseline values
Fasting glucose concentrations | From baseline to week 4
  Plasma fasting glucose concentrations at week 4 adjusting for baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Bath, United Kingdom